CLINICAL TRIAL: NCT01431495
Title: Clinical Assessment of Pidogrel® Versus Plavix®
Brief Title: Clinical Assessment of Pidogrel® Versus Plavix® (CAPP)
Acronym: (CAPP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPP-study
Record Dates: First submitted 2011-08-25; First posted 2011-09-09 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Coronary Disease
Keywords: platelet agregation; clopidogrel; major adverse cardiac events (MACE)
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- plavix (Active Comparator): patient treated by the princeps
  Interventions: Drug: Plavix
- Pidogrel (Active Comparator): patient treated by Pidogrel
  Interventions: Drug: Pidogrel

INTERVENTIONS:
Drug: Pidogrel — Pidogrel(R)75 mg/day for period ranging from 1 to 6 months.
  Arms: Pidogrel
Drug: Plavix — Plavix(R) 75 mg/day for period ranging from 1 to 6 months.
  Arms: plavix

SUMMARY:
This study aims to demonstrate non-inferiority of Pidogrel ® compared to Plavix ® in patients with coronary disease:

* Primary Outcome Measures: measure of platelet reactivity by VerifyNow assay after 600 mg loading dose or after the last maintenance dose (75 mg).
* Secondary Outcome Measures: Time to first occurrence of major cardio-vascular events (MACE).
* Safety Criteria: severe bleeding (GUSTO scale).

DETAILED DESCRIPTION:
after randomization of patients in both groups (Plavix or Pidogrel), the measure of platelet activity by the VerifyNow assay, 4 to 12 hours after the loading dose of 600mg or after the last dose of clopidogrel for patients on maintenance dose. The VerifyNow assay will determine: - The PRU:-P2Y12 Reaction Units-

-% Of platelet inhibition It will be considered low responder or clopidogrel resistant patient with PRU> 235 or %inhibition <15%.

Monitoring of patients included in the study will take place over a period of 12 months, MACE will be notified and dated. MACE criteria are: angina, myocardial infarction, coronary angioplasty, coronary artery bypass graft, and stroke.

Each hemorrhagic event will be notified and classified according to the GUSTO scale.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,
* Old (e) over 20 years
* Patients hospitalized for acute coronary syndrome (Whatever the T and troponin)
* Patients with proven coronary candidates for treatment with clopidogrel (who received a loading dose of 600mg over 2 hours and treated with 75mg / d of clopidogrel for longer than 7 days)

Exclusion Criteria:

* Patients unwilling.
* Patient participating in another study.
* Patients with cardiogenic shock
* Patient on anti GpIIbIIIa or stopped less than 72 hours before the test aggregability
* Patients scheduled for surgery in less than 6 months.
* Patients candidates for coronary angioplasty
* Patients who underwent TAC + / - bare stent fewer than 30 days.
* Patients who underwent stenting with ATC active there is less than 12 months.
* ischemic stroke older than 6 weeks.
* History of hemorrhagic stroke (any time)
* Patients on warfarin or candidates
* Patients with a different anti ADP (ticlopidine, prasugrel)
* Patients with indication for clopidogrel-cons (side effects, bleeding ...)
* Thrombocytopenia <100000/mm3
* anemia (Ht <30%)
* Thrombocythaemia (Ht> 52%)
* Patients seeking treatment for an elective forms of Clopidogrel.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
- study the respective effects of Pidogrel ® and Plavix ® on platelet aggregation through the test VerifyNow ® - Time to first occurrence of post-randomization major adverse cardiac events (MACE) | 06 months

CONTACTS AND LOCATIONS:
Overall Officials: Rachid MECHMECHE, MD, Study Chair — hospital La RABTA
Locations (1):
- cardiology department, hospital La RABTA, Tunis, Tunis BAB Souika, Tunisia